CLINICAL TRIAL: NCT00238238
Title: A Randomized Phase II Trial of Rituximab Versus Lenalidomide (REVLIMID™, Cc-5013) (IND#73034) Versus Rituximab + Lenalidomide in Recurrent Follicular Non-Hodgkin Lymphoma (NHL) That is Not Rituximab-Refractory
Brief Title: Rituximab and/or Lenalidomide in Treating Patients With Follicular Non-Hodgkin's Lymphoma That is Not Refractory to Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50401; CALGB-50401; U10CA031946 (NIH); CDR0000442872 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I - rituximab (Active Comparator): Patients receive rituximab IV on days 1, 8, 15, and 22.
  Interventions: Biological: rituximab
- Arm II - lenalidomide (Experimental): Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide
- Arm III - lenalidomide and rituximab (Experimental): Patients receive lenalidomide as in arm II. Patients also receive rituximab IV on days 8, 15, 22 and 29.
  Interventions: Biological: rituximab; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — Given IV
  Arms: Arm I - rituximab; Arm III - lenalidomide and rituximab
Drug: lenalidomide — Given orally
  Arms: Arm II - lenalidomide; Arm III - lenalidomide and rituximab

SUMMARY:
Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Lenalidomide may also stop the growth of non-Hodgkin's lymphoma by blocking blood flow to the cancer. Giving rituximab together with lenalidomide may kill more cancer cells. This randomized phase II trial is studying how well rituximab and/or lenalidomide work in treating patients with follicular non-Hodgkin's lymphoma that is not refractory to rituximab.

DETAILED DESCRIPTION:
Outline:

This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms. Please see the "Arms" section for a description of each treatment arm. The primary and secondary objectives of the study are provided below.

Primary Objectives:

* To determine the response rate (overall and complete) after lenalidomide therapy and rituximab + lenalidomide in follicular NHL patients who have relapsed.
* To determine time to progression after lenalidomide therapy and rituximab and lenalidomide in follicular NHL patients who have relapsed.

Secondary Objectives:

* To compare the time to progression of the previous rituximab regimen to that obtained subsequently to lenalidomide therapy and rituximab + lenalidomide.
* To determine the toxicity profile of lenalidomide therapy and of rituximab and lenalidomide in follicular NHL patients who have received a previous rituximab regimen.
* To correlate Fc receptor polymorphism profiling with response to lenalidomide or rituximab + lenalidomide in previously treated patients with follicular NHL who have relapsed.
* To evaluate changes in Natural Killer (NK) cells, activated NK cells, activated T-cells and several plasma cytokines followed by rituximab therapy and correlation of observed changes to objective response rates.

After completion of study treatment, patients are followed for up to 10 years from study entry.

ELIGIBILITY:
* Documentation of Disease

  * Previously treated, histologically confirmed follicle center cell lymphoma, World Health Organization (WHO) classification, grade 1, 2, or 3a
  * Institutional flow cytometry or immunohistochemistry must confirm Cluster of Differentiation 20 (CD20) antigen expression.
* Prior Treatment

  * Patient must have been treated with rituximab either alone or in combination with chemotherapy.
  * Patient must have a time to progression of ≥ 6 months from last rituximab dose.
  * No corticosteroids within two weeks prior to study, except for maintenance therapy for a non-malignant disease. Maintenance therapy dose may not exceed 20 mg/day prednisone or equivalent.
  * No prior radioimmunotherapy within 12 months of study entry.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Measurable disease must be present either on physical examination or imaging studies. Non-measurable disease alone is not acceptable. Any tumor mass >1 cm is acceptable.Lesions that are considered non-measurable include the following:

  * Bone lesions
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Bone marrow
* No known Central Nervous System (CNS) involvement by lymphoma.
* No known Human Immunodeficiency Virus (HIV) infection.
* Non-pregnant and non-nursing.
* Patients with a "currently active" second malignancy, other than non-melanoma skin cancers, are not eligible.
* Patients with a recent history (within 3 months of study entry) of Deep Vein Thrombosis/Pulmonary Embolism (DVT/PE) are not eligible.
* Required Initial Laboratory Values:

  * Absolute Neutrophil Count (ANC) ≥ 1000/µL
  * Platelet count ≥ 75,000/µL
  * Creatinine < 1.5 x Upper Limit of Normal (ULN) unless attributed to lymphoma or calculated clearance > 50 mL/min (patients on dialysis are not eligible)
  * Total Bilirubin ≤ 2 x ULN unless attributed to lymphoma or Gilbert's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-03; Primary Completion 2012-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Leonard, MD, Study Chair — Weill Medical College of Cornell University
Locations (79):
- United States (79):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Leonard JP, Jung SH, Johnson J, Pitcher BN, Bartlett NL, Blum KA, Czuczman M, Giguere JK, Cheson BD. Randomized Trial of Lenalidomide Alone Versus Lenalidomide Plus Rituximab in Patients With Recurrent Follicular Lymphoma: CALGB 50401 (Alliance). J Clin Oncol. 2015 Nov 1;33(31):3635-40. doi: 10.1200/JCO.2014.59.9258. Epub 2015 Aug 24. PMID 26304886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2006 and April 2011, 97 participants were accrued to the study.
Pre-assignment Details: Three participants assigned to the lenalidomide arm alone arm never began treatment, and the rituximab arm was discontinued early.
Groups:
- Arm I - Rituximab: Patients receive rituximab 375 mg/m^2 IV on days 1, 8, 15, and 22.
- Arm II - Lenalidomide: Patients receive oral lenalidomide 15 mg once daily on days 1-21 in cycle 1, then 20 mg once daily on days 1-21 cycle 2-12. Treatment repeats every 28 days.
- Arm III - Lenalidomide and Rituximab: Patients receive oral lenalidomide 15 mg once daily on days 1-21 in cycle 1, then 20 mg once daily on days 1-21 cycle 2-12 Patients also receive rituximab 375 mg/m^2 IV on days 8, 15, 22 and 29.
Period: Overall Study
Arm/Group | Arm I - Rituximab | Arm II - Lenalidomide | Arm III - Lenalidomide and Rituximab
Started | 3 | 48 | 46
Completed | 3 | 45 | 46
Not Completed | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Three participants assigned to the lenalidomide arm alone arm never began treatment. Participants on the rituximab arm was discontinued early; in order to avoid potential identification of patients, no results will be entered for this arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Rituximab | Arm II - Lenalidomide | Arm III - Lenalidomide and Rituximab | Total
Number analyzed (Participants) | 0 | 45 | 46 | 91
Age, Continuous [Median (Full Range); unit: years] |  | 63 [34 to 85] | 64 [36 to 89] | 63 [34 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 18 | 19 | 37
  Male |  | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0
  Asian |  | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander |  | 1 | 0 | 1
  Black or African American |  | 3 | 1 | 4
  White |  | 37 | 44 | 81
  More than one race |  | 0 | 0 | 0
  Unknown or Not Reported |  | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States |  | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response is assessed by investigator according to International Working Group (IWG) criteria. A complete response requires disappearance of all evidence of disease. A partial response is a >/= 50% decrease in the sum of products of 6 largest dominant nodes or nodal masses as well as for splenic and hepatic nodules. No increase in size of nodes, liver or spleen and no new sites of disease.
Time Frame: Duration of treatment (12 cycles)
Population: Three participants assigned to the lenalidomide arm alone arm never began treatment, and the rituximab arm was discontinued early.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I - Rituximab | Arm II - Lenalidomide | Arm III - Lenalidomide and Rituximab
Number analyzed (Participants) | 0 | 45 | 46
percentage of participants |  | 53.3 [37.9 to 68.3] | 76.1 [61.2 to 87.4]
Statistical Analysis 1: Comparison: Arm II - Lenalidomide vs Arm III - Lenalidomide and Rituximab; Test type: Superiority or Other; p = 0.29, Fisher Exact

2. Primary Outcome: Time to Progression
Description: Time to progression (TTP) is defined as the time from study entry until progression or death without progression. The median TTP with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Up to 10 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I - Rituximab | Arm II - Lenalidomide | Arm III - Lenalidomide and Rituximab
Number analyzed (Participants) | 0 | 45 | 46
years |  | 1.1 [0.8 to 1.2] | 2 [1.7 to 3.0]
Statistical Analysis 1: Comparison: Arm II - Lenalidomide vs Arm III - Lenalidomide and Rituximab; Test type: Superiority or Other; p = 0.002, Log Rank

ADVERSE EVENTS:
Description: 90 participants, on Arms II and III, were evaluable for adverse events.
Arm/Group | Arm I - Rituximab | Arm II - Lenalidomide | Arm III - Lenalidomide and Rituximab
Serious Adverse Events (participants affected / at risk) | 0/0 | 8/45 | 12/45
Other Adverse Events (participants affected / at risk) | 0/0 | 44/45 | 41/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Rituximab (N=0) | Arm II - Lenalidomide (N=45) | Arm III - Lenalidomide and Rituximab (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 4 (4)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (4)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (8)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 5 (6) | 7 (11)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (4)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 4 (4) | 5 (6)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 4 (6)
Platelet count decreased (Investigations) | 0 (0) | 6 (7) | 5 (6)
Weight loss (Investigations) | 0 (0) | 2 (2) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Kidney pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Rituximab (N=0) | Arm II - Lenalidomide (N=45) | Arm III - Lenalidomide and Rituximab (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 19 (89) | 17 (86)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 6 (24)
Dry eye syndrome (Eye disorders) | 0 (0) | 3 (5) | 2 (3)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (3) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (6) | 4 (9)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 21 (40) | 16 (45)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 14 (46) | 14 (34)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (12) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (7) | 2 (4)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Gastroscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 16 (40) | 12 (32)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (9) | 6 (7)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (7)
Chills (General disorders) | 0 (0) | 2 (2) | 7 (7)
Edema limbs (General disorders) | 0 (0) | 9 (28) | 6 (11)
Fatigue (General disorders) | 0 (0) | 35 (138) | 33 (166)
Fever (General disorders) | 0 (0) | 2 (2) | 7 (7)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 4 (5) | 4 (16)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 12 (12)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (4) | 3 (3)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 8 (15)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 5 (7) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (11)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (5) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 8 (27) | 9 (35)
Alkaline phosphatase increased (Investigations) | 0 (0) | 5 (14) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 8 (21) | 10 (33)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (6) | 8 (31)
Creatinine increased (Investigations) | 0 (0) | 6 (10) | 4 (14)
INR increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (3) | 2 (15)
Leukocyte count decreased (Investigations) | 0 (0) | 21 (86) | 16 (131)
Lymphocyte count decreased (Investigations) | 0 (0) | 9 (21) | 13 (80)
Neutrophil count decreased (Investigations) | 0 (0) | 19 (94) | 25 (123)
Platelet count decreased (Investigations) | 0 (0) | 25 (96) | 23 (114)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight loss (Investigations) | 0 (0) | 2 (2) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 6 (12) | 5 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 15 (50) | 14 (55)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 7 (12) | 6 (18)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 8 (24) | 10 (38)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (11)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 7 (14)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 6 (10) | 6 (23)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 7 (13) | 6 (27)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 6 (20) | 6 (16)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 7 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (9) | 6 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 3 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 4 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (16) | 6 (20)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 4 (9)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 8 (11) | 10 (16)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (18) | 3 (7)
Headache (Nervous system disorders) | 0 (0) | 5 (16) | 5 (10)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 15 (32) | 17 (51)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 4 (15) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (6) | 4 (10)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (7)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (20) | 6 (12)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (15) | 11 (30)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (13) | 8 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 4 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (7)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (12) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (15) | 8 (22)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (17) | 6 (16)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (16) | 10 (13)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (9) | 8 (11)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (8) | 3 (4)
Hot flashes (Vascular disorders) | 0 (0) | 1 (8) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (5) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 4 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less